CLINICAL TRIAL: NCT05976178
Title: Descriptive, Prospective Study of the Characteristics of Chronic Pain in Patients With Addiction to at Least One Substance
Brief Title: Study of the Characteristics of Chronic Pain in Patients With Addiction
Acronym: ADDICTALGO
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Responsible Party: Principal Investigator, Alexandre Cauchie, Principal Investigator, Groupe Hospitalier de Bretagne Sud
Other Study IDs: 56LORC_2021_ADDICTALGO
Record Dates: First submitted 2023-07-11; First posted 2023-08-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Addiction
MeSH Terms: conditions — Chronic Pain; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
It is described in the literature a higher prevalence of pain in patients with an addiction but there are few studies describing the pain profile of patients with use disorder.

Pain has a very negative impact on the quality of life of opioid substituted patients. Improving knowledge on this point would make it possible to better guide specific care.

The investigator proposes to conduct a single-center descriptive observational study using questionnaires, without changing the management of patients with chronic pain.

The primary objective of the study is to determine the prevalence of chronic pain in patients with substance addiction hospitalized for addiction treatment.

DETAILED DESCRIPTION:
It is described in the literature a higher prevalence of pain in patients with an addiction but there are few studies describing the pain profile of patients with use disorder.

Pain has a very negative impact on the quality of life of opioid substituted patients. Improving knowledge on this point would make it possible to better guide specific care.

The investigator proposes to conduct a single-center descriptive observational study using questionnaires, without changing the management of patients with chronic pain. All patients admitted to hospitalization in the addiction department of the LORIENT Hospital will be offered participation in the study.

The primary objective of the study is to determine the prevalence of chronic pain in patients with substance addiction hospitalized for addiction treatment.

The study will also evaluate the impact on daily activities of the presence of two chronic pathologies: chronic pain and addiction, describe the frequency of the two main psychiatric comorbidities of chronic pain: anxiety and depression, describe the different components of chronic pain in patients with substance addiction, and get information on analgesic medications.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Presence of addiction to at least one substance, based on DSM-5 criteria
* Hospitalized in the addiction service of LORIENT Hospital
* Knowing how to read and write French
* Not objecting to their participation in the study after informed information

Exclusion Criteria:

* Already included during a precedent hospitalization
* Adults subject to legal protection or deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the addictology department of LORIENT Hospital, in full hospitalization or in a day hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic pain in patients with substance addiction hospitalized for addiction treatment. | During the hospitalization, maximum 1 month
  Percentage of patients presenting with pain for more than three months among patients hospitalized in an addiction service for the management of an addiction

SECONDARY OUTCOMES:
Pain intensity in the last 24 hours | During the hospitalization, maximum 1 month
  Results of the Brief Pain Inventory : worst and least of pain in the last 24 hours
Interference of pain on the quality of life | During the hospitalization, maximum 1 month
  Result of Brief pain inventory on general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. On a scale from 0 (does not interfere) to 10 (completely interferes)
Localisation of pain | During the hospitalization, maximum 1 month
  Drawing on a diagram of a human body
Describe the frequency of the two main psychiatric comorbidities of chronic pain: anxiety | During the hospitalization, maximum 1 month
  Results of the anxiety scale of Hospital Anxiety and Depression scale. Positive if > 8. Minimum 0, maximum 21
Describe the frequency of the two main psychiatric comorbidities of chronic pain: depression | During the hospitalization, maximum 1 month
  Results of the depression scale of Hospital Anxiety and Depression scale. Positive if > 8. Minimum 0, maximum 21
Describe the prevalence of fibromyalgia among patients with substance addiction | During the hospitalization, maximum 1 month
  Results of the Fibromyalgia Rapid Screening Tool. Suspicion of fibromyalgia if >5 yes. Maximum 6 yes
Information on analgesics medication | During the hospitalization, maximum 1 month
  Collection of current analgesic medication taken every day
Describe the prevalence of neuropathic pain among patients with substance addiction | During the hospitalization, maximum 1 month
  Results of the DN3 (neuropathic pain 3). Suspicion of neuropathic pain when > 3/7

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Cauchie, MD, Principal Investigator — GH Bretagne Sud
Locations (1):
- Groupe Hospitalier Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenblum A, Joseph H, Fong C, Kipnis S, Cleland C, Portenoy RK. Prevalence and characteristics of chronic pain among chemically dependent patients in methadone maintenance and residential treatment facilities. JAMA. 2003 May 14;289(18):2370-8. doi: 10.1001/jama.289.18.2370. PMID 12746360
- [Background] Lusted A, Roerecke M, Goldner E, Rehm J, Fischer B. Prevalence of pain among nonmedical prescription opioid users in substance use treatment populations: systematic review and meta-analyses. Pain Physician. 2013 Nov-Dec;16(6):E671-84. PMID 24284850
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Voon P, Greer AM, Amlani A, Newman C, Burmeister C, Buxton JA. Pain as a risk factor for substance use: a qualitative study of people who use drugs in British Columbia, Canada. Harm Reduct J. 2018 Jul 5;15(1):35. doi: 10.1186/s12954-018-0241-y. PMID 29976203
- [Background] Larson MJ, Paasche-Orlow M, Cheng DM, Lloyd-Travaglini C, Saitz R, Samet JH. Persistent pain is associated with substance use after detoxification: a prospective cohort analysis. Addiction. 2007 May;102(5):752-60. doi: 10.1111/j.1360-0443.2007.01759.x. PMID 17506152